CLINICAL TRIAL: NCT02374619
Title: The Effect of Eccentric Exercise and Iron Supplementation on Blood Redox Status and Muscle Performance in Different Age Groups
Brief Title: Iron Supplementation and Eccentric Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Athanasios Z. Jamurtas, Associate Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: UTH2010
Record Dates: First submitted 2015-02-16; First posted 2015-03-02 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Muscle Damage; Oxidative Stress
Keywords: eccentric exercise; pro-oxidants; free radicals; adults; children

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iron supplement (Experimental): Oral supplementation
  Interventions: Dietary Supplement: Iron supplement Resoferon Ferrous Sulfate
- Control (Placebo Comparator): Oral supplementation
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Iron supplement Resoferon Ferrous Sulfate — Oral supplementation with one tablet of iron supplement [Resoferon Ferrous Sulfate 125 (37) mg]
  Arms: Iron supplement
Dietary Supplement: Placebo
  Arms: Control

SUMMARY:
Iron supplementation is very common in athletes, probably due to its catalytic role on the oxygen transport and optimal function of oxidative enzymes and proteins during exercise.

Iron is also characterized as a potent pro-oxidant, as it can lead to increased production of reactive oxygen and nitrogen species (RONS) that are involved in critical biological processes, such as gene expression, signal transduction and enzyme activity. In exercise, low levels of RONS are essential for optimal force production, whereas excessive production of RONS can cause contractile dysfunction, resulting in muscle weakness and fatigue. On the other hand, RONS are involved in signaling pathways and up-regulation of the expression of several genes, and therefore, RONS can provoke favorable effects such as training adaptations.

The purpose of the present study is to investigate the effect of iron supplementation on redox status, muscle damage and muscle performance after an acute bout of a valid muscle damaging eccentric exercise model in adults and children.

DETAILED DESCRIPTION:
Eccentric muscle work is an essential part of human daily activities, such as walking, and in particular, when walking downhill or descending stairs. It is also a component of almost all of the athletic actions. The most notable and well-described effect of eccentric exercise is the muscle damage that peaks one to three days after exercise and is accompanied by several hematological, biochemical and physiological responses. Excessive production of reactive oxygen and nitrogen species (RONS) has been reported as a result of eccentric exercise. The typical approach so far, was to provide antioxidants to minimize oxidative stress, yet the effectiveness of such an approach is still under debate. Earlier studies reported positive effects of antioxidant supplementation on muscle performance, muscle damage and redox status, whereas more recently, well-received studies pointed towards the negative impact of antioxidant supplementation.

Iron is an essential element for the completion of numerous important biological functions, and also for optimal exercise performance. It is a vital component for the formation of oxygen-transport and iron-storage proteins hemoglobin and myoglobin, and for the most favorable function of many oxidative enzymes that affect the intracellular metabolism. Therefore, iron supplementation is commonly used to avoid exercise-induced perturbations of iron homeostasis and maintain the required iron stores that are necessary to address exercise needs or enhance physical performance. Iron is also characterized as a potent pro-oxidant, as it can lead to increased production of reactive oxygen and nitrogen species (RONS) that are involved in critical biological processes, such as gene expression, signal transduction and enzyme activity. Nevertheless, the role of iron on modifying redox responses after eccentric exercise has not yet been examined.

In a double blind, randomized cross over study that will be conducted in two cycles, healthy men and boys will receive either the iron supplement (37mg of elemental iron per day for three weeks before and one week after the eccentric exercise) or the placebo.

Blood samples will be collected: a) in adults prior to, at the end of first supplementation period, 24, 48,72 and 96 hours following an acute bout of eccentric exercise (5 sets x 15 max reps), and b) in children prior to, at the end of first supplementation period and 72 hours following the same exercise protocol. Blood drawings will be repeated at the same time points during the second supplementation cycle.

The aims of the present research are to investigate:

* The effect of an acute bout of eccentric exercise on muscle performance, redox status, and iron status.
* The effect of three weeks of iron supplementation on muscle performance, redox status, and iron status.
* The effect of four weeks of iron supplementation on muscle damage, muscle performance, and redox status after an acute eccentric exercise bout.
* The effect of age on muscle damage, muscle performance and redox status after an acute eccentric exercise bout and iron supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Physiological body mass index (BMI).
* Physiological health profile.
* Subject provides written informed consent.

Exclusion Criteria:

* Professional athlete.
* Consumed any nutritional supplement the last 3 months.
* Performed pure eccentric exercise the last 6 months.
* Non Caucasian.

Ages: 10 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2011-12; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Changes in Maximum isometric torque (N.m) | Before the beginning of iron supplementation (baseline) at the end of the first supplementation period (3 weeks: pre-eccentric exercise), immediately after the eccentric exercise, and 24 hours, 48 hours, 72 hours, 96 hours after the eccentric exercise
  An isokinetic dynamometer (Cybex, Ronkonkoma, NY) will be used for the estimation of changes in isometric knee extensor's peak torque at 90o knee flexion between baseline and after 3 weeks of supplementation (pre-eccentric exercise), and also between pre-eccentric exercise and 24 hours, 48 hours, 72 hours, 96 hours after the eccentric exercise. The average of the three best maximal voluntary contractions with the subjects' one lower extremity will be recorded. To ensure that the subjects provide their maximal effort, the measurements will be repeated if the difference between the lower and the higher torque value exceed 10%. There will be two minutes rest between isometric efforts.
Changes in Maximum concentric torque (N.m) | Before the beginning of iron supplementation (baseline) at the end of the first supplementation period (3 weeks: pre-eccentric exercise), immediately after the eccentric exercise, and 24 hours, 48 hours, 72 hours, 96 hours after the eccentric exercise
  An isokinetic dynamometer (Cybex, Ronkonkoma, NY) will be used for the estimation of changes in isokinetic knee extensor's peak torque at 60o/sec angular velocity between baseline and after 3 weeks of supplementation (pre-eccentric exercise), and also between pre-eccentric exercise and 24 hours, 48 hours, 72 hours, 96 hours after the eccentric exercise. The higher absolute value of five maximal voluntary contractions with the subjects' one lower extremity will be recorded.
Changes in Maximum eccentric torque (N.m) | Before the beginning of iron supplementation (baseline) at the end of the first supplementation period (3 weeks: pre-eccentric exercise), immediately after the eccentric exercise, and 24 hours, 48 hours, 72 hours, 96 hours after the eccentric exercise
  An isokinetic dynamometer (Cybex, Ronkonkoma, NY) will be used for the estimation of changes in isokinetic knee extensor's peak torque at 60o/sec angular velocity between baseline and after 3 weeks of supplementation (pre-eccentric exercise), and also between pre-eccentric exercise and 24 hours, 48 hours, 72 hours, 96 hours after the eccentric exercise. The higher absolute value of five maximal voluntary contractions with the subjects' one lower extremity will be recorded.
Changes in Range of motion, ROM (degrees) | Before the beginning of iron supplementation (baseline) at the end of the first supplementation period (3 weeks: pre-eccentric exercise), immediately after the eccentric exercise, and 24 hours, 48 hours, 72 hours, 96 hours after the eccentric exercise
  The assessment of changes in pain-free ROM between baseline and after 3 weeks of supplementation (pre-eccentric exercise), and also between pre-eccentric exercise and 24 hours, 48 hours, 72 hours, 96 hours after the eccentric exercise, will be performed manually using the isokinetic dynamometer. The investigator will move the calf at a very low angular velocity from 0 knee extension to the position where the subject will feel any discomfort.
Changes in Delayed onset muscle soreness, DOMS (scale 1-10) | Before the beginning of iron supplementation (baseline) at the end of the first supplementation period (3 weeks: pre-eccentric exercise), immediately after the eccentric exercise, and 24 hours, 48 hours, 72 hours, 96 hours after the eccentric exercise
  Each participant will assess changes in delayed onset of muscle soreness (DOMS) during walking and squat movement (90o knee flexion) and perceived soreness between baseline and after 3 weeks of supplementation (pre-eccentric exercise), and also between pre-eccentric exercise and 24 hours, 48 hours, 72 hours, 96 hours after the eccentric exercise. DOMS and perceived soreness will be rated on a scale ranging from 1 (normal) to 10 (very sore).
Changes in Creatine kinase, CK (activity IU) | Before the beginning of iron supplementation (baseline), at the end of the first supplementation period (3 weeks: pre exercise), and 72h after the eccentric exercise
  CK activity will be measured as a general indicator of muscle damage. Changes in CK activity between baseline and after 3 weeks of supplementation (pre-eccentric exercise), and also between pre-eccentric exercise and 24 hours, 48 hours, 72 hours, 96 hours after the eccentric exercise will be estimated in a Clinical Chemistry Analyzer Z1145 (Zafiropoulos Diagnostica, Athens, Greece) with commercially available kits (Zafiropoulos, Athens, Greece).

SECONDARY OUTCOMES:
Changes in Reduced glutathione, GSH (μmol/g Hb) | Adults: at baseline, pre-eccentric exercise, 24,48,72 & 96 hours after the eccentric exercise. Children: at baseline, pre-eccentric exercise and 72 hours after the eccentric exercise
  GSH will be measured as a general index of oxidative stress. Changes in GSH between baseline and after 3 weeks of supplementation (pre-eccentric exercise), and also between pre-eccentric exercise and 24 hours, 48 hours, 72 hours, 96 hours after the eccentric exercise will be assessed. For GSH, 20 μL of erythrocyte lysate will be treated with 5% TCA mixed with 660 μL of 67 mM sodium potassium phosphate (pH 8.0) and 330 ΜL of 1 mM 5,5-dithiobis-2 nitrobenzoate. The samples will be incubated in the dark at room temperature for 45 min, and the absorbance will be read at 412 nm.
Changes in Oxidized glutathione, GSSG (μmol/g Hb) | Adults: at baseline, pre-eccentric exercise, 24,48,72 & 96 hours after the eccentric exercise. Children: at baseline, pre-eccentric exercise and 72 hours after the eccentric exercise
  GSSG will be measured as a general index of oxidative stress. Changes in GSSG between baseline and after 3 weeks of supplementation (pre-eccentric exercise), and also between pre-eccentric exercise and 24 hours, 48 hours, 72 hours, 96 hours after the eccentric exercise will be investigated. GSSG will be assayed by treating 50 μL of erythrocyte lysate with 5% TCA and neutralized up to pH 7.0-7.5. One microliter of 2-vinylpyridine will be added, and the samples will be incubated for 2 h. Sample will be treated with TCA and will be mixed with 600 μL of 143 mM sodium phosphate 100 ΜL of 3 mM NADPH, 100 ΜL of 10 mM 5,5-dithiobis-2-nitrobenzoate, and 194 μL of distilled water. After the addition of 1 μL of glutathione reductase, the change in absorbance at 412 nm will be read for 3 min.
Changes in Thiobarbituric acid-reactive substances, TBARS (μM) | Adults: at baseline, pre-eccentric exercise, 24,48,72 & 96 hours after the eccentric exercise. Children: at baseline, pre-eccentric exercise and 72 hours after the eccentric exercise
  TBARS will be measured as an index of lipid peroxidation. Changes in TBARS between baseline and after 3 weeks of supplementation (pre-eccentric exercise), and also between pre-eccentric exercise and 24 hours, 48 hours, 72 hours, 96 hours after the eccentric exercise will be investigated. For TBARS determination, 100 μL of plasma will be mixed with 500 ΜL of 35% TCA and 500 μL of Tris-HCl (200 mM, pH 7.4) and will be incubated for 10 min at room temperature. One milliliter of 2 M Na2SO4 and 55 mM thiobarbituric acid solution will be added, and the samples will be incubated at 95O C for 45 min. The samples will be cooled on ice for 5 min and then will be vortexed after adding 1 mL of 70% TCA. The samples will be centrifuged at 15,000g for 3 min, and the absorbance of the supernatant will be read at 530 nm.
Changes in Protein carbonyls, PC (nmol/mg pr) | Adults: at baseline, pre-eccentric exercise, 24,48,72 & 96 hours after the eccentric exercise. Children: at baseline, pre-eccentric exercise and 72 hours after the eccentric exercise
  Carbonyls will be measured as an index of protein oxidation. Changes in PC between baseline and after 3 weeks of supplementation (pre-eccentric exercise), and also between pre-eccentric exercise and 24 hours, 48 hours, 72 hours, 96 hours after the eccentric exercise will be investigated. Protein carbonyls will be determined adding 50 μL of 20% TCA to 50 μL of plasma. Samples will be incubated in the dark at room temperature for 1 hour. The supernatant will be discarded, and 1 mL of 10% TCA will be added. The supernatant will be discarded, and 1 mL of ethanol-ethyl acetate will be added and centrifuged. The supernatant will be discarded, and 1 mL of 5 M urea will be added, vortexed, and incubated at 37C for 15 min. The samples will be centrifuged at 15,000g for 3 min at 4C, and the absorbance will be read at 375 nm.
Changes in Catalase (μmol/min/mg Hb) | Adults: at baseline, pre-eccentric exercise, 24,48,72 & 96 hours after the eccentric exercise. Children: at baseline, pre-eccentric exercise and 72 hours after the eccentric exercise
  Catalase will be measured as one of the main antioxidant enzyme of erythrocytes. Changes in catalase between baseline and after 3 weeks of supplementation (pre-eccentric exercise), and also between pre-eccentric exercise and 24 hours, 48 hours, 72 hours, 96 hours after the eccentric exercise will be investigated. Catalase activity will be determined adding 4 μL of erythrocyte lysate, 2955 μL of 67 mM sodium potassium phosphate (pH 7.4), and the samples will be incubated at 37C for 10 min. Five microliters of 30% hydrogen peroxide was added to the samples, and the change in absorbance will immediately read at 240 nm for 1.5 min.
Changes in Total antioxidant capacity, TAC (mm DPPH) | Adults: at baseline, pre-eccentric exercise, 24,48,72 & 96 hours after the eccentric exercise. Children: at baseline, pre-eccentric exercise and 72 hours after the eccentric exercise
  Changes in TAC between baseline and after 3 weeks of supplementation (pre-eccentric exercise), and also between pre-eccentric exercise and 24 hours, 48 hours, 72 hours, 96 hours after the eccentric exercise will be investigated. TAC will be determined adding 20 μL of plasma to 480 ΜL of 10 mM sodium potassium phosphate (pH 7.4) and 500 μL of 0.1 mM 2,2-diphenyl-1-picrylhydrazyl (DPPH) free radical, and the samples will be incubated in the dark for 30 min at room temperature. The samples will be centrifuged for 3 min at 20,000g, and the absorbance will be read at 520 nm.
Changes in Uric acid (μm) | Adults: at baseline, pre-eccentric exercise, 24,48,72 & 96 hours after the eccentric exercise. Children: at baseline, pre-eccentric exercise and 72 hours after the eccentric exercise
  Uric acid will be measured as the main antioxidant component of blood plasma. Changes in Uric acid between baseline and after 3 weeks of supplementation (pre-eccentric exercise), and also between pre-eccentric exercise and 24 hours, 48 hours, 72 hours, 96 hours after the eccentric exercise will be investigated. It will be measured in a Clinical Chemistry Analyzer Z1145 (Zafiropoulos Diagnostica, Athens, Greece) with commercially available kits (Zafiropoulos, Athens, Greece).
Changes in Bilirubin (μM) | Adults: at baseline, pre-eccentric exercise, 24,48,72 & 96 hours after the eccentric exercise. Children: at baseline, pre-eccentric exercise and 72 hours after the eccentric exercise
  Changes in Bilirubin between baseline and after 3 weeks of supplementation (pre-eccentric exercise), and also between pre-eccentric exercise and 24 hours, 48 hours, 72 hours, 96 hours after the eccentric exercise will be investigated. Bilirubin will be measured in a Clinical Chemistry Analyzer Z1145 (Zafiropoulos Diagnostica, Athens, Greece) with commercially available kits (Zafiropoulos, Athens, Greece).
Changes in Iron concentration (mg/dL) | Adults: at baseline, pre-eccentric exercise, 24,48,72 & 96 hours after the eccentric exercise. Children: at baseline, pre-eccentric exercise and 72 hours after the eccentric exercise
  Changes in Iron concentration between baseline and after 3 weeks of supplementation (pre-eccentric exercise), and also between pre-eccentric exercise and 24 hours, 48 hours, 72 hours, 96 hours after the eccentric exercise will be investigated. Iron concentration will be measured in a Clinical Chemistry Analyzer Z1145 (Zafiropoulos Diagnostica, Athens, Greece) with commercially available kits (Zafiropoulos, Athens, Greece).
Changes in Total Iron Binding Capacity (TIBC) (μmol/L) | Adults: at baseline, pre-eccentric exercise, 24,48,72 & 96 hours after the eccentric exercise. Children: at baseline, pre-eccentric exercise and 72 hours after the eccentric exercise
  Changes in TIBC between baseline and after 3 weeks of supplementation (pre-eccentric exercise), and also between pre-eccentric exercise and 24 hours, 48 hours, 72 hours, 96 hours after the eccentric exercise will be investigated. TIBC will be measured in a Clinical Chemistry Analyzer Z1145 (Zafiropoulos Diagnostica, Athens, Greece) with commercially available kits (Zafiropoulos, Athens, Greece).
Changes in Transferin saturation (TS) (%) | Adults: at baseline, pre-eccentric exercise, 24,48,72 & 96 hours after the eccentric exercise. Children: at baseline, pre-eccentric exercise and 72 hours after the eccentric exercise
  Changes in TS between baseline and after 3 weeks of supplementation (pre-eccentric exercise), and also between pre-eccentric exercise and 24 hours, 48 hours, 72 hours, 96 hours after the eccentric exercise will be investigated. Transferrin saturation will be calculated from iron and TIBC values.
Changes in Ferritin (ng/mL) | Adults: at baseline, pre-eccentric exercise, 24,48,72 & 96 hours after the eccentric exercise. Children: at baseline, pre-eccentric exercise and 72 hours after the eccentric exercise
  Changes in Ferritin concentration between baseline and after 3 weeks of supplementation (pre-eccentric exercise), and also between pre-eccentric exercise and 24 hours, 48 hours, 72 hours, 96 hours after the eccentric exercise will be investigated. For the determination of serum Ferritin an immunoenzymometric assay (EIA) kit based on sandwich ELISA will be used (Accubind, Monobind Inc., USA®) which contains all the necessary reagents. The absorbance in each well will be read at 450nm using a microplate reader (Biochrom Asys Expert 96, UK). For the calculation of the concentration of ferritin, a dose response curve was used according to the assay directions.

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios Z Jamurtas, Dr, Study Chair — University of Thessaly

REFERENCES:
- [Background] Theodorou AA, Nikolaidis MG, Paschalis V, Koutsias S, Panayiotou G, Fatouros IG, Koutedakis Y, Jamurtas AZ. No effect of antioxidant supplementation on muscle performance and blood redox status adaptations to eccentric training. Am J Clin Nutr. 2011 Jun;93(6):1373-83. doi: 10.3945/ajcn.110.009266. Epub 2011 Apr 20. PMID 21508092
- [Background] Gomez-Cabrera MC, Martinez A, Santangelo G, Pallardo FV, Sastre J, Vina J. Oxidative stress in marathon runners: interest of antioxidant supplementation. Br J Nutr. 2006 Aug;96 Suppl 1:S31-3. doi: 10.1079/bjn20061696. PMID 16923247
- [Derived] Deli CK, Fatouros IG, Paschalis V, Tsiokanos A, Georgakouli K, Zalavras A, Avloniti A, Koutedakis Y, Jamurtas AZ. Iron Supplementation Effects on Redox Status following Aseptic Skeletal Muscle Trauma in Adults and Children. Oxid Med Cell Longev. 2017;2017:4120421. doi: 10.1155/2017/4120421. Epub 2017 Jan 22. PMID 28203319